CLINICAL TRIAL: NCT05563753
Title: Impact of Early Antibiotic Therapy on Vaccination Response in Preterm Infants
Brief Title: Early Antibiotic Therapy and Vaccinations in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 024/2022BO1
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Vaccination Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool samples for microbiome analyses blood for vaccination titers and b- and t-cell analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ABT in the first week of life: VLBWI with gestational age between 24+0 and 31+6 weeks of gestation with antibiotic treatment in the first week of life
  Interventions: Drug: ABT
- no antibiotic therapy (ABT) in the first week of life: VLBWI with gestational age between 24+0 and 31+6 weeks of gestation without antibiotic treatment in the first week of life

INTERVENTIONS:
Drug: ABT — any antibiotic therapy in the first week of life
  Other Names: any antibiotic therapy
  Groups: ABT in the first week of life

SUMMARY:
Since the neonatal sepsis is still one of the most common causes of death in preterm infants up to 80% receive an perinatal antibiotic treatment. It is also known that an antibiotic treatment is one of the most important influences for the establishment of the intestinal microbiome. This again is important for the development of an healthy neonatal immunosystem. A pilot study showed that an antibiotic therapy in the first week of life had a negative influence on the vaccine titers of preterm infants.

In this study it will be further investigated if an early antibiotic treatment influences the development of the adaptive immunosystem in preterm infants and if this antibiotic treatment effects the development of the intestinal microbiome.

DETAILED DESCRIPTION:
The study wants to investigate the impact of the antibiotic treatment in the first week of live on the adaptive immunosystem. For this the antibody titers against Hepatitis B, Poliomyelitis, Pertussis, Haemophilus influenzae B, Tetanus, Diphtheria and Pneumococcus of very low birth weight infants (VLBWI) who receive an early antibiotic therapy will be compared with the antibody titers of infants who did not receive antibiotic treatment. Further the development of b- and t-cells will be tested.

To show the modulation of the intestinal microbiome through antibiotics stool samples of VLBWI with and without antibiotic therapy in first week of life will be tested for their composition and diversity as well as for the production of short-chained fatty acids (SCFA) In this study 82 VLBWI (42 per group) will be included. Infants will be matched by age and gender.

ELIGIBILITY:
Inclusion Criteria:

* born at University Hospital Tübingen
* received at least one dose of antibiotics during the first week of life

Exclusion Criteria:

* genetic disorders
* chronic infections
* hematological disorders
* treatment with immunoglobulins during the first 60 days of life
* immunological disorders
* infants with Hepatitis B positive mothers

Ages: 24 Weeks to 32 Weeks | Sex: All
Age Groups: Child
Study Population: Preterm infants with a gestational age between 24+0 and 31+6 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Vaccination response | 7 Month
  Measurement of antibody titers against Hepatitis B, Poliomyelitis, Pertussis, Haemophilus Influenzae B, Tetanus, Diphteria and Pneumococcus four month after the first received vaccination
Analyses of b- and t-cells development | 7 Month
  Analyses of b- and t-cell development with the adjusted age of 4 moth

SECONDARY OUTCOMES:
Microbiome analyses | 7 Month
  Analyses of the microbiome composition at the age of 14 days and adjusted age of 4 month
Analyses of SCFA production of the intestinal microbiome | 7 month
  Analyses of SCFA production of the intestinal microbiome with the age of corrected 4 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospial Tübingen, Tübingen, Baden-Wurttemberg, Germany